CLINICAL TRIAL: NCT06712329
Title: Chronic Plantar Fasciitis: Which is More Effective? Prolotherapy/Extracorporeal Shock Wave Therapy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayşe Ukbe Baykut, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACHBİLKENTAUBAYKUT001
Record Dates: First submitted 2024-11-16; First posted 2024-12-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Plantar Fasciitis
Keywords: prolotherapy; extracorporeal shock wave therapy; plantar pressure distribution; plantar fascia thickness
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Extracorporeal Shockwave Therapy; Prolotherapy

STUDY DESIGN:
Intervention Model Description: 1. Inceler Medical, Modus Focused ESWT
  2. 15% dextrose solution injection
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- extracorporeal shock wave therapy group (Experimental): In the ESWT group, a total of 1800 to 2000 focused shock waves (0.15-0.25 mJ/mm² sessions with a frequency of 3-4 Hz) were applied
  Interventions: Other: extracorporeal shock wave therapy
- Prolotherapy Group (Experimental): The prolotherapy group was administered a 3-ml injection of a 15% dextrose solution.
  Interventions: Other: Prolotherapy

INTERVENTIONS:
Other: extracorporeal shock wave therapy — ESWT (Inceler Medical, Modus Focused ESWT, Turkey) was conducted by a single investigator in accordance with a standardised protocol. The patients were positioned prone on the examination table, with the affected limb placed in a supported position. The focused shockwave was applied in a circular motion along the insertion site of the plantar fascia and over the plantar fascia itself. The participants received 1,800 to 2,000 focused shock waves (0.15-0.25 mJ/mm² session with a frequency of 3-4 Hz). The frequency of the pulses was increased in a gradual manner, in accordance with the maximum tolerable degree of pain for each patient. A minimum dose of 1,000 mJ/mm² was administered. The ESWT was conducted in three sessions, with a two-week interval between each session.
  Other Names: eswt
  Arms: extracorporeal shock wave therapy group
Other: Prolotherapy — The solution employed for dextrose prolotherapy comprised 1.5 ml of 30% dextrose and 1.5 ml of 0.9% isotonic sodium chloride solution, resulting in a total of 3 ml of 15% dextrose solution. . All procedures were conducted by the same investigator. A dextrose solution was infused into the centre and around the damaged area using a peppering technique. Following the procedure, patients were advised to remain in a supine position with their feet restrained for a period of 15 minutes.. Prolotherapy was repeated on three occasions, with each session occurring at a two-week interval
  Other Names: dextrose prolotherapy
  Arms: Prolotherapy Group

SUMMARY:
The primary objective of this prospective study was to compare the effects of ESWT (extracorporeal shock wave therapy ) and prolotherapy on pain and foot function in patients with chronic plantar fasciitis. In addition, the study was to investigate the changes in plantar pressure distribution and plantar fascia thickness measured by ultrasonography after ESWT and prolotherapy.

The fundamental questions that investigators want to answer are as follows:

[question 1]:Do ESWT and prolotherapy improve pain and foot function in patients with chronic plantar fasciitis? [question 2]:Do ESWT and prolotherapy change plantar pressure distribution and plantar fascia thickness in patients with chronic plantar fasciitis?

DETAILED DESCRIPTION:
Chronic plantar fasciitis is a prevalent musculoskeletal disorder that results in discomfort and impaired functionality within the plantar surface of the foot. In instances where conservative treatment proves ineffective, it can complicate the management of the condition. Two invasive treatment options, namely extracorporeal shock wave therapy (ESWT) and prolotherapy, are available for the management of plantar fasciitis, with the objective of providing pain and functional improvement. The objective of this study was to compare the effects of ESWT and prolotherapy on pain, foot function, plantar fascia thickness and plantar pressure distribution in patients with chronic plantar fasciitis.

A total of 70 patients who did not respond to conservative treatment were included in this prospective, randomised controlled study. Following a clinical and ultrasonographic evaluation, the patients were randomly assigned to one of two groups. The study population was divided into two groups: the ESWT group (n = 36) and the prolotherapy group (n = 34). In the ESWT group, a total of 1800 to 2000 focused shock waves (0.15-0.25 mJ/mm² sessions with a frequency of 3-4 Hz) were applied. The prolotherapy group was administered a 3-ml injection of a 15% dextrose solution. The ESWT and prolotherapy treatments were administered in a total of three sessions, with two-week intervals between each session. The efficacy of the treatment was evaluated using a number of different measures, including the Visual Analogue Scale (VAS), the Foot and Ankle Ability Measurement (FAAM), the thickness of the plantar fascia and the distribution of plantar pressure. The evaluations were conducted at the outset of the study, at the six-week mark, and at the 12-week mark following the final intervention.

ELIGIBILITY:
Inclusion Criteria:

1. participants must be aged between 18 and 75 years
2. they must have experienced heel pain for a period of at least three months
3. they must exhibit pain and tenderness upon palpation of the medial aspect of the calcaneal tuberosity with the ankle in full dorsiflexion
4. they must have demonstrated no response to conservative treatment for a minimum of three months.

In cases where symptoms were present on both sides, the more prominent side was included.

Exclusion Criteria:

1. Inflammatory rheumatic disease
2. Dermatological lesion on the heel
3. Pregnancy
4. Infection
5. Malignancy
6. Coagulopathy
7. Pacemaker
8. Peripheral circulatory disorder
9. A neurological disorder, such as radiculopathy or polyneuropathy
10. Previous ESWT, dextrose prolotherapy, or surgical procedure to the heel region
11. A local corticosteroid injection or oral corticosteroids in the last six weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) | baseline - 6th week-12th week
  The Visual Analogue Scale (VAS) was employed to evaluate the general perception of pain and the pain experienced at the first step upon rising. The scale ranges from 0 to 10, with a score of 0 indicating no pain and a score of 10 indicating the most severe pain imaginable

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | baseline - 6th week-12th week
  The Foot and Ankle Ability Measure (FAAM) was developed to assess the physical function of individuals with foot pathology. FAAM is a self-administered questionnaire consisting of 29 items, 21 of which pertain to activities of daily living (ADL) and 8 to sports. Each item of the FAAM is scored on a 5-point Likert scale with 4 points representing no difficulty at all; 3 points, slight difficulty; 2 points, moderate difficulty; 1 point, extreme difficulty; and 0 points, unable to do. The sixth option is not applicable if patients feel that this item does not concern them. If all items are answered, the ADL and sports subscales have a maximum score of 84 and 32, respectively. The obtained scores are transformed to percentages by dividing them with the maximum potential score and then multiplying the result by 100. A high score in both categories is indicative of a high level of physical functioning
Thickness of the plantar fascia | baseline - 6th week-12th week
  A high-resolution ultrasound (5-13 MHz linear transducer, LOGIQ 9; GE Healthcare, China) was employed to ascertain the thickness of the plantar fascia. Ultrasonography measurements were conducted by the same individual, who has over five years of experience in this field. The participants were positioned in a prone manner with their ankles maintained in a neutral position. The thickness was measured in a vertical direction, commencing from the hyperechogenic border of the calcaneus bone and continuing until it reached the lower hyperechogenic edge of the plantar fascia. An average of three plantar fascia thickness measurements were taken at each assessment to minimise potential errors. The plantar fascia thickness was evaluated by a physiatrist who was unaware of the treatment groups
Plantar pressure distribution | baseline - 6th week-12th week
  All participants underwent a static plantar pressure distribution assessment utilising the Formetric 4D system (DIERS MedicalSystems, Germany). In the test, each participant was required to stand on the platform, barefoot, with their feet side by side and facing forward for a period of five seconds. The parameters subjected to analysis were hindfoot plantar pressure (percent) and forefoot plantar pressure (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe U Baykut, Principal Investigator — Ankara Şehir Hastanesi Bilkent
Locations (1):
- Ankara Şehir Hastanesi Bilkent, Ankara, çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
all collected IPD

REFERENCES:
- See also: Pub Med — https://pubmed.ncbi.nlm.nih.gov/